CLINICAL TRIAL: NCT03693703
Title: Cost-efficacy of a Preliminary Diagnostic Program Using Bi-parametric Magnetic Resonance Imaging in Men With Suspicion of Prostate Cancer and no Previous Prostate Biopsy: a Prospective Randomized Clinical Study Comparing Multiparametric and Bi-parametric Magnetic Resonance Imaging Results
Brief Title: Comparison of Multi-parametric and Bi-parametric Magnetic Resonance Imaging in Men With Suspicion of Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: bpMRscr16
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Prostatic Neoplasm
Keywords: magnetic resonance imaging; prostate biopsy; microRNA
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bi-parametric MRI (Experimental): Patients will undergo axial T2-weighted and diffusion-weighted imaging (no contrast agent injection)
  Interventions: Diagnostic Test: bi-parametric MRI
- multi-parametric MRI (Active Comparator): Patients will undergo multiparametric MRI including morphological study (T2- and T1-weighted imaging) and functional acquisitions (diffusion-weighted and dynamic contrast-enhanced imaging)
  Interventions: Diagnostic Test: multi-parametric MRI

INTERVENTIONS:
Diagnostic Test: bi-parametric MRI — Axial T2-weighted and diffusion-weighted imaging with no endorectal coil nor intravenous contrast agent administration
  Arms: bi-parametric MRI
Diagnostic Test: multi-parametric MRI — T2-weighted imaging in the three planes, diffusion-weighted and dynamic contrast-enhanced imaging using endorectal coil and intravenous contrast agent administration
  Arms: multi-parametric MRI

SUMMARY:
To compare the detection rate of biparametric (bp) magnetic resonance imaging (MRI) for clinically significant prostate cancer (PCa) with that of multiparametric (mp)-MRI, in biopsy-naïve patients. Today, bp-MRI is not the standard diagnostic procedure, however preliminary studies showed its non-inferiority with respect to mp-MRI. Its implementation on a wide scale could significantly reduce examination costs (no iv contrast agent and no endorectal coil), and study time.

Secondary objectives will be:

* to assess specificity of a blood test based on microRNA (miR) score in biopsy-naïve patients, using pathological assessment after MR-guided biopsy as reference standard. If specificity of the miR score is higher than that of PSA, then fewer patients will undergo unnecessary MRI, thus increasing the efficiency of the diagnostic pipeline for PCa;
* to develop a clinical decision support system (CDSS) based on MRI and circulating miR evaluation, to stratify patients according to their risk of PCa progression, using pathological assessment after prostatectomy as reference standard. Patients will be stratified into two classes of risk: i) low-risk PCa, in which patients may benefit from a conservative approach (i.e. active surveillance), and ii) medium/high-risk PCa in which patients should undergo radical treatment (i.e. surgery or radiation therapy).

DETAILED DESCRIPTION:
The trial is a prospective, randomized, two-arms study with a 2:1 ratio. Subjects meeting the inclusion criteria will be randomized either into the bp-MRI group (arm A), or the mp-MRI one (arm B). All subjects will perform blood sampling in EDTA tubes before undergoing imaging session. Plasma will be isolated within 1 hour from sampling, with a double round centrifugation, aliquoted and stored at -80°C before undergoing miR analysis.

MRI will be performed with a 1.5 T using axial T2w and diffusion-weighted imaging for subjects in arm A with no endorectal coil and no intravenous contrast agent. Men randomized in arm B will undergo MRI with T2w in the three acquisition planes, diffusion-weighted and dynamic contrast-enhanced imaging usign endorectal coil.

Random biopsy will be performed in subjects with no suspicious regions for PCa found on MRI. Men with suspicious regions on MRI will be invited to a targeted or in-bore biopsy.

ELIGIBILITY:
Inclusion Criteria:

* age <= 75 years
* PSA <= 15 ng/ml
* no previous prostate biopsy
* negative digital rectal examination
* signed infomed conset

Exclusion Criteria:

* known prostate cancer diagnosis
* previous prostate biopsy or surgery
* contraindication to MRI
* non-cooperative subjects

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Detection rate of bi-parametric MRI, and of mp-MRI in men at risk for PCa and with no previous prostate biopsy | 3 months
  Sensitivity, specificity, PPV and NPV will be measured

SECONDARY OUTCOMES:
Dimension of lesions identified at bp-MRI/mp-MRI; | 2 weeks
  Mean lesion dimension will be assessed in each study arm
The proportion of clinically significant PCa identified at bp-MRI; | 2 weeks
  The number of clinically significant PCa over the total number of PCa detected at bp-MRI will be measured
Positive predictive value of miR test alone and in combination with PSA blood test in identifying histologically confirmed PCa patients | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Russo, MD, Principal Investigator — Fondazione del Piemonte per l'Oncologia
Locations (1):
- Fondazione del Piemonte per l'Oncologia - Candiolo Cancer Institute, Candiolo, Turin, Italy

REFERENCES:
- [Derived] Russo F, Mazzetti S, Regge D, Ambrosini I, Giannini V, Manfredi M, De Luca S, Bollito E, Porpiglia F. Diagnostic Accuracy of Single-plane Biparametric and Multiparametric Magnetic Resonance Imaging in Prostate Cancer: A Randomized Noninferiority Trial in Biopsy-naive Men. Eur Urol Oncol. 2021 Dec;4(6):855-862. doi: 10.1016/j.euo.2021.03.007. Epub 2021 Apr 21. PMID 33893066